CLINICAL TRIAL: NCT04470154
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial Evaluating the Safety, Pharmacokinetics, and Efficacy of HSK21542 Injection in Subjects Undergoing Hemodialysis
Brief Title: A Study Evaluating the Safety, Pharmacokinetics, and Efficacy of HSK21542 Injection in Subjects Undergoing Hemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK21542-203
Record Dates: First submitted 2020-07-07; First posted 2020-07-14 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Uremic Pruritus

STUDY DESIGN:
Intervention Model Description: This study is a multicenter study, which is divided into two stages. The first stage is a dose escalation, randomized, double-blind, placebo-controlled study of multiple intravenous administration within one week in hemodialysis subjects. The second stage is a randomized, double-blind, placebo-controlled study of Administration for 12 weeks in hemodialysis subjects with moderate or severe pruritus.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Stage I: 0.05 μg/kg (Experimental): IV HSK21542 0.05 μg/kg solution（active or placebo） administered after each dialysis session within 2h±30 min (3 times/week).
  Interventions: Drug: Stage I:HSK21542 0.05 μg/kg
- Stage I: 0.15 μg/kg (Experimental): IV HSK21542 0.15 μg/kg solution（active or placebo） administered after each dialysis session within 2h±30 min (3 times/week).
  Interventions: Drug: Stage I:HSK21542 0.15 μg/kg
- Stage I: 0.30 μg/kg (Experimental): IV HSK21542 0.30 μg/kg solution（active or placebo） administered after each dialysis session within 2h±30 min (3 times/week).
  Interventions: Drug: Stage I:HSK21542 0.30 μg/kg
- Stage I: 0.80 μg/kg (Experimental): IV HSK21542 0.80 μg/kg solution（active or placebo） administered after each dialysis session within 2h±30 min (3 times/week).
  Interventions: Drug: Stage I:HSK21542 0.80 μg/kg
- Stage II: 0.3 μg/kg (Experimental): IV HSK21542 0.3 μg/kg solution（active or placebo） administered after each dialysis session within 10 min (3 times/week).
  Interventions: Drug: Stage II:HSK21542 0.3 μg/kg
- Stage II: 0.6 μg/kg (Experimental): IV HSK21542 0.3 μg/kg solution（active or placebo） administered after each dialysis session within 10 min (3 times/week).
  Interventions: Drug: Stage II:HSK21542 0.6 μg/kg

INTERVENTIONS:
Drug: Stage I:HSK21542 0.05 μg/kg — Following the principle of dose escalation and starting from the low dose of 0.05 μg/kg to the high dose 0.80 μg/kg
  Arms: Stage I: 0.05 μg/kg
Drug: Stage I:HSK21542 0.15 μg/kg — Following the principle of dose escalation and starting from the low dose of 0.05 μg/kg to the high dose 0.80 μg/kg
  Arms: Stage I: 0.15 μg/kg
Drug: Stage I:HSK21542 0.30 μg/kg — Following the principle of dose escalation and starting from the low dose of 0.05 μg/kg to the high dose 0.80 μg/kg
  Arms: Stage I: 0.30 μg/kg
Drug: Stage I:HSK21542 0.80 μg/kg — Following the principle of dose escalation and starting from the low dose of 0.05 μg/kg to the high dose 0.80 μg/kg
  Arms: Stage I: 0.80 μg/kg
Drug: Stage II:HSK21542 0.3 μg/kg — Randomized to HSK21542 0.3 μg/kg or 0.6 μg/kg or the corresponding placebo group
  Arms: Stage II: 0.3 μg/kg
Drug: Stage II:HSK21542 0.6 μg/kg — Randomized to HSK21542 0.3 μg/kg or 0.6 μg/kg or the corresponding placebo group
  Arms: Stage II: 0.6 μg/kg

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled phase II clinical trial. The main objective is to evaluate the safety, pharmacokinetics, and efficacy of HSK21542 injection in subjects undergoing hemodialysis

DETAILED DESCRIPTION:
This study is a multicenter study, which is divided into two stages. The first stage is a dose escalation, randomized, double-blind, placebo-controlled study of multiple intravenous administration within one week in hemodialysis subjects. The second stage is a randomized, double-blind, placebo-controlled study of Administration for 12 weeks in hemodialysis subjects with moderate or severe pruritus. In the second stage, consist of a Screening Visit, a 7-day Run-in Period, a 12 week Double-blind Treatment Period, and a 2-week Discontinuation Period. Informed consent will be obtained prior to performing any study-specific procedures. The Screening Visit will occur within 8 to 28 days prior to randomization to assess eligibility.

ELIGIBILITY:
Stage1: Inclusion Criteria:

1. Subjects who are willing to sign an informed consent form, fully understand the objectives and purposes of the study, and are willing to comply with the study protocol before any of the study-related procedures start;
2. Aged ≥ 18 and ≤ 75 years old, male or female;
3. Dry weight ≥ 50.0 kg at screening, body mass index (BMI = weight (kg) / height2 [m2]) in the range of 16.0-30.0 kg/m^2 (inclusive);
4. Patients with end-stage renal diseases who receive hemodialysis (including hemodiafiltration) 3 times in a week prior to screening for at least 3 months;
5. Patients with at least two occurrences of single-compartment urea clearance (sp Kt/V, see Appendix 7 for the calculation formula) ≥ 1.2, or at least two occurrences of urea reduction ratio (URR) ≥ 65%, or one occurrence of sp Kt/V ≥ 1.2 and one occurrence of URR ≥ 65% on different days of dialysis within 3 months before screening;
6. Male subjects must agree to use condoms in sexual intercourse during the study and within 3 months after the last dose; female subjects should have had menopause for at least one year, or should have had permanent sterilization (e.g., fallopian tube occlusion, hysterectomy, bilateral salpingectomy); or women of childbearing potential must agree to take effective contraceptive measures during the study and within 3 months after the last dose, such as oral contraceptives, condoms, and contraceptive films.

Stage1: Exclusion Criteria:

1. Expected to undergo kidney transplantation and/or parathyroidectomy during the study;
2. History of allergy to opioids, such as urticaria (Note: adverse effects related to opioid use, such as constipation and nausea, are not included as the exclusion criteria in this study);
3. Used opioids within one week before screening, or unable to avoid the use of opioids other than the investigational product during the study;
4. Participated in any clinical trial of other drug or medical device within 1 month before screening (received study medication or treated by the medical device in the clinical trial);
5. Used blood perfusion within 3 months before screening;
6. History of medication or drug abuse;
7. Average daily alcohol consumption greater than 15 g (15 g of alcohol is equivalent to 450 mL of beer or 150 mL of wine or 50 mL of light liquor) within 3 months before screening;
8. Unable to comply with the standard dietary plan and unable to avoid coffee or tea during the study;
9. Blood pressure of upper limbs in the supine position at screening: systolic blood pressure < 90 mmHg, or diastolic blood pressure < 60 mmHg, or systolic blood pressure > 180 mmHg, or diastolic blood pressure > 110 mmHg;
10. New York Heart Association (NYHA) Class ≥ III at screening; or confirmed to have abnormal ECG at screening and determined by the investigator to be inappropriate to be enrolled, including QTcF ≥ 480 ms;
11. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or total bilirubin ≥ 1.5 × upper limit of normal (ULN) at screening;
12. Blood sodium > 155 mmol/L at screening;
13. Hemoglobin ≤ 80 g/L at screening;
14. Positive for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), syphilis antibody, or human immunodeficiency virus (HIV) antibody at screening;
15. Underwent major surgery (determined by the investigator as major surgery) within 3 months before screening;
16. Having a total blood loss of ≥ 200mL within 1 month before screening, except for the blood loss during menstruation in females;
17. Females who are pregnant or breastfeeding;
18. Any physiological or psychological diseases or conditions that may increase the risk of the trial, affect the subject's compliance with the protocol, or affect the subject's completion of the trial, as judged by the study physician, including but not limited to:

    1. Severe mental illness or cognitive impairment (e.g., dementia);
    2. Any other relevant acute or chronic neurological and psychiatric diseases (e.g., encephalopathy, coma, delirium) within 3 months before screening;
    3. Patients with malignant tumors (including malignant tumors that have been cured without recurrence).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Stage I：Safety of HSK21542 injection for multiple times within one week in hemodialysis subjects | From screening up to D14
  Adverse events (AEs) and serious adverse events (SAEs)，Vital signs、Physical examination, Laboratory examination, ECG
Stage II：At week 12, the change in weekly average of daily Worst Itch NRS (WI-NRS) from baseline in subjects undergoing hemodialysis | 12 week
  Change from baseline in average NRS score of itch at week 12

SECONDARY OUTCOMES:
Stage I：Area under the plasma concentration versus time curve (AUC) | 1 week
  Plasma HSK21542 Area Under the Concentration-time Curve (AUC)
Stage I：Time to the peak plasma concentration (Tmax) | 1 week
  Time to Maximum Plasma HSK21542 Concentration
Stage I：Maximum Concentration (Cmax) | 1 week
  Maximum Concentration of HSK21542
Stage I：Half-time (T1/2) | 1 week
  Half-time of HSK21542
Stage I：Total body clearance following intravenous administration (CL) | 1 week
  Total body clearance following intravenous administration of HSK21542
Stage I：Volume of distribution following intravenous administration (Vss) | 1 week
  Volume of distribution following intravenous administration of HSK21542
Stage I：trough concentration (Cmin) | 1 week
  trough concentration of HSK21542
Stage I：Change from baseline in average daily Worst Itch NRS (WI-NRS) and Itch-related Quality of Life as Assessed by Skindex-16 Scale Score | 1 week
  Intensity of itch will be measured using an NRS used to indicate the intensity of the worst itching over the past 24 hours using a 0 to 10 numeric rating scale, where "0" represents "no itching" and "10" represents "worst itching imaginable".
  The Skindex-16 Scale is a multidimensional questionnaire which assesses itch-related quality of life over the past week. The questions cover 3 domains: disease, mood/emotional distress, and social functioning domain. The Skindex-16 has 16 questions; the total Skindex-16 score ranges from 0 to 100. A higher total score represents worse quality of life.
Stage I：Correlation between prolactin level and drug exposure of HSK21542 injection in hemodialysis subjects | 1 week
  Detect prolactin concentration before and after administration
Stage II: Safety of HSK21542 injection in the treatment of moderate and severe pruritus in hemodialysis subjects for 12 weeks | 12 weeks
  Adverse events (AEs) and serious adverse events (SAEs)，Vital signs、Physical examination, Laboratory examination, ECG
Stage II：Area under the plasma concentration versus time curve (AUC) | 12 weeks
  Plasma Area Under the Concentration-time Curve of HSK21542
Stage II：Time to Maximum plasma concentration (Tmax) | 12 weeks
  Time to Maximum Plasma Concentration of HSK21542
Stage II：Maximum Concentration (Cmax) | 12 weeks
  Maximum Concentration of HSK21542
Stage II：Half-time (T1/2) | 12 weeks
  Half-time (T1/2) of HSK21542
Stage II：Total body clearance following intravenous administration (CL) | 12 weeks
  Total body clearance following intravenous administration of HSK21542
Stage II：Volume of distribution following intravenous administration (Vss) | 12 weeks
  Volume of distribution following intravenous administration of HSK21542
Stage II: The proportion of subjects change from baseline ≥3 points with respect to the weekly mean of the daily 24-hour Worst Itching Intensity NRS Score at Week 12 | 12 week
  Intensity of itch will be measured using an NRS used to indicate the intensity of the worst itching over the past 24 hours using a 0 to 10 numeric rating scale, where "0" represents "no itching" and "10" represents "worst itching imaginable". LS means estimated percent, odds ratio and P value used logistic and Log-binomial regression model.
Stage II: The proportion of subjects change from baseline ≥4 points with respect to the weekly mean of the daily 24-hour Worst Itching Intensity NRS Score at Week 12 | 12 week
  Intensity of itch will be measured using an NRS used to indicate the intensity of the worst itching over the past 24 hours using a 0 to 10 numeric rating scale, where "0" represents "no itching" and "10" represents "worst itching imaginable". LS means estimated percent, odds ratio and P value used logistic and Log-binomial regression model.
Stage II：Change from baseline in Itch-related Quality of Life as Assessed by Skindex-16 and 5-D Scale Score | 12 week
  The Skindex-16 Scale is a multidimensional questionnaire which assesses itch-related quality of life over the past week. The questions cover 3 domains: disease, mood/emotional distress, and social functioning domain. The Skindex-16 has 16 questions; the total Skindex-16 score ranges from 0 to 100. A higher total score represents worse quality of life.
  The 5-D Itch Scale is a multidimensional questionnaire which assesses itch-related quality of life over the past 2 weeks. The questions cover five dimensions of itch including the duration of itch/day, degree, direction (improvement/worsening), disability (impact on activities such as work), and body distribution of itch. The 5-D Itch Scale has 5 questions; the total 5-D Itch Scale score ranges from 5 to 25, with higher scores indicating worse responses.
Stage II: Weekly mean value of the daily 24-hour Worst Itching Intensity NRS Score within 2 weeks after drug withdrawal after 12 weeks of administration | 14 week
  Intensity of itch will be measured using an NRS used to indicate the intensity of the worst itching over the past 24 hours using a 0 to 10 numeric rating scale, where "0" represents "no itching" and "10" represents "worst itching imaginable".
Stage II: Weekly mean value of the ShOWS and OOWS Score within 2 weeks after drug withdrawal after 12 weeks of administration | 14 week
  According to the weekly mean of ShOWS and OOWS scores, combined with AE, comprehensively evaluate whether there is drug withdrawal reaction.
Stage II: Change from baseline in the level of serum IL-6，IL-31，TNF-α，and hs-CRP | 12 weeks
  Evaluate the effect of HSK21542 on IL-6, IL-31, TNF- α and hs-CRP levels.
Stage II: Change from baseline in the level of serum iPTH | 12 weeks
  Evaluate the effect of HSK21542 on iPTH levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Guizhou Medical University Affiliated Hospital, Guiyang, Guizhou, China

REFERENCES:
- [Derived] Pan M, Wang G, Zhou L, Xu Y, Yao L, Wu C, Mei C, Zhao Z, Sun D, Guan T, Chen Q, Shi M, Xu H, Zeng W, Li F, Yan R, Liu BC. Safety and effectiveness of HSK21542 for hemodialysis patients: a multiple ascending dose study. Front Pharmacol. 2023 Oct 9;14:1203642. doi: 10.3389/fphar.2023.1203642. eCollection 2023. PMID 37876731